CLINICAL TRIAL: NCT05618002
Title: Lemborexant vs Zopiclone vs Clonidine for Insomnia Treatment in Chronic Pain Patients
Status: Recruiting | Type: Observational
Sponsor: Salem Anaesthesia Pain Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: SalemAnaesth2022 LemborexZop
Record Dates: First submitted 2022-11-08; First posted 2022-11-16 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Chronic Insomnia; Chronic Pain
Keywords: Sedative; Hypnotic
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Chronic Pain | interventions — lemborexant; zopiclone; Clonidine

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Lemborexant — For insomnia treatment, each patient ingests Lemborexant or Zopiclone or Clonidine on alternate nights. Each patient uses a special validated sleep diary to collect data.
  Other Names: Zopiclone; Clonidine

SUMMARY:
Prospective observational crossover study of 150 consenting adult patients who are undergoing chronic pain management. For insomnia treatment, each patient ingests prescribed doses of Lemborexant or Zopiclone or Clonidine on alternate nights. Each patient uses a special validated sleep diary to collect data including pain score, sleep score, sleep duration, sleep medication type, and adverse effects. Each patient completes the diary for 3 continuous weeks. Pain is measured using the numeric pain rating scale. Sleep score is measured using the Likert sleep scale. A change in the pain or sleep scores by 2-points is considered significant.

DETAILED DESCRIPTION:
Objectives: Chronic pain is usually associated with insomnia. The objective of this clinical study is to compare the safety and efficacy of Lemborexant or Zopiclone or Clonidine; for the management of chronic insomnia in patients with chronic pain.

Methods: Prospective observational crossover study of 150 consenting adult patients who are undergoing chronic pain management. For insomnia treatment, each patient ingests prescribed doses of Lemborexant or Zopiclone or Clonidine on alternate nights. Each patient uses a special validated sleep diary to collect data including pain score, sleep score, sleep duration, sleep medication type, and adverse effects. Each patient completes the diary for 3 continuous weeks. Pain is measured using the numeric pain rating scale. Sleep score is measured using the Likert sleep scale. A change in the pain or sleep scores by 2-points is considered significant. Data analyzed with IBM® SPSS® Statistics 25 (IBM Corp, Armonk, NY); using Student's t-test, ANOVA, Pearson Chi-square test, and regression analysis. P-value <0.05 is considered significant.

ELIGIBILITY:
Inclusion Criteria:

* adult chronic pain patients
* good treatment compliance
* severe chronic insomnia
* failure of non-pharmacologic sleep therapy
* regular zopiclone therapy for 3 months or more
* regular sleep diary
* regular pain diary
* informed consent for diary review
* consent for clinical record quality assurance review

Exclusion Criteria:

* obstructive sleep apnoea
* body mass index (BMI) ≥40
* organ insufficiency
* cognitive disorder
* inability to provide consent
* major neuropsychiatric disorder
* unreliable diary
* cannabis use
* regular alcohol intake
* stimulant use
* substance abuse
* poor treatment compliance
* high dose opioid
* gabapentinoid use
* sedative use
* mild insomina
* irregular zopiclone intake
* regular zopiclone therapy for less than 3 months
* previous adverse/allergic reactions to clonidine or zopiclone

Ages: 20 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult chronic pain clinic patients who have severe chronic insomnia; and undergoing medication treatment for insomnia.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-11-08 (Actual); Primary Completion 2025-12-11 (Estimated); Study Completion 2025-12-11 (Estimated)

PRIMARY OUTCOMES:
Sleep quality score, objective measurement using the validated Likert sleep scale | 3 weeks
  Sleep quality score, using the Likert sleep scale of 0 to 10, low scores indicate poor sleep, high scores indicate better sleep

SECONDARY OUTCOMES:
Pain score, objective measurement using the validated Numeric Pain Rating scale | 3 weeks
  Pain score, using the Numeric Pain Rating scale of 0 to 10, low scores indicate less pain, high scores indicate worse pain

CONTACTS AND LOCATIONS:
Overall Officials: Olu Bamgbade, MD,FRCPC, Principal Investigator — Salem Anaesthesia Pain Clinic
Locations (1):
- Salem Anaesthesia Pain Clinic, Surrey, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bamgbade OA, Tai-Osagbemi J, Bamgbade DO, Murphy-Akpieyi O, Fadire A, Soni NK, Mumporeze L. Clonidine is better than zopiclone for insomnia treatment in chronic pain patients. J Clin Sleep Med. 2022 Jun 1;18(6):1565-1571. doi: 10.5664/jcsm.9930. PMID 35112665